CLINICAL TRIAL: NCT05037760
Title: A Phase 2 Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of KER-050 as Monotherapy or in Combination With Ruxolitinib in Participants With Myelofibrosis
Brief Title: A Study of Elritercept Alone or Together With Ruxolitinib in Adults With Myelofibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KER050-MF-301; 2023-507468-38-00 (EU CTIS Number)
Record Dates: First submitted 2021-08-23; First posted 2021-09-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Myelofibrosis
Keywords: Thrombocytopenia; Anemia; Red blood cells; Bone marrow; KER-050; drug therapy; elritercept
MeSH Terms: conditions — Primary Myelofibrosis; Thrombocytopenia; Anemia | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm 1A: Elritercept (Experimental): Participants with anemia who have discontinued Janus Kinase (JAK) inhibitor(s) or are intolerant or ineligible for JAK inhibitor(s) will be administered escalating doses of elritercept, starting at 0.75 milligrams per kilograms (mg/kg) followed by 1.5 mg/kg and 4.5 mg/kg subcutaneously (SC), every 4 weeks for 13 cycles for a total Treatment Period of 52 weeks. Each cycle is 28 days.
  Interventions: Drug: Elritercept
- Arm 1B: Elritercept + Ruxolitinib (Experimental): Participants with anemia who have been receiving ruxolitinib for ≥8 weeks prior to Cycle 1 Day 1 (C1D1) and are on a stable dose for ≥4 weeks prior to C1D1 will be administered escalating doses of elritercept, starting at 0.75 mg/kg and followed by 1.5 mg/kg and 4.5 mg/kg, SC, every 4 weeks for 13 cycles in combination with ruxolitinib therapy for a total Treatment Period of 52 weeks. Each cycle is 28 days.
  Interventions: Drug: Elritercept; Drug: Ruxolitinib
- Arm 2A: Elritercept (Experimental): Participants with with anemia who have discontinued JAK inhibitor(s) or are intolerant or ineligible for JAK inhibitor(s) will be administered elritercept, 3.75 mg/kg, SC, every 4 weeks for 13 cycles for a total Treatment Period of 52 weeks. Each cycle is 28 days.
  Interventions: Drug: Elritercept
- Arm 2B: Elritercept + Ruxolitinib (Experimental): Participants with anemia who have been receiving ruxolitinib for ≥8 weeks prior to C1D1 and are on a stable dose for ≥4 weeks prior to C1D1 will be administered elritercept, 3.75 mg/kg, SC, every 4 weeks for 13 cycles in combination with ruxolitinib therapy for a total Treatment Period of 52 weeks. Each cycle is 28 days.
  Interventions: Drug: Elritercept; Drug: Ruxolitinib
- Experimental: Arm 2C: Elritercept (Brazil Only) (Experimental): Participants from Brazil with anemia who have received no prior treatment with JAK inhibitor(s) and have no access to JAK inhibitor therapy will be administered elritercept, 3.75 mg/kg, SC, every 4 weeks for 13 cycles for a total Treatment Period of 52 weeks. Each cycle is 28 days.
  Interventions: Drug: Elritercept
- Long-Term Extension (Experimental): Participants from Arms 1A, 1B, 2A, 2B and 2C benefiting from the continued elritercept treatment as a monotherapy or in combination with ruxolitinib can continue to receive elritercept in this long-term extension phase until elritercept becomes commercially available or until elritercept is no longer being developed for the treatment of MF.
  Interventions: Drug: Elritercept; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Elritercept — Elritercept SC injection.
  Other Names: KER-050; TAK-226
Drug: Ruxolitinib — Ruxolitinib tablet.
  Arms: Arm 1B: Elritercept + Ruxolitinib; Arm 2B: Elritercept + Ruxolitinib; Long-Term Extension

SUMMARY:
The main aim of this study is to learn how safe elritercept is and how well it is tolerated when taken alone and in combination with the JAK inhibitor, ruxolitinib. Other aims are to learn about the effects of elritercept on the signs and symptoms of MF when taken with or without ruxolitinib and to learn how elritercept affects the body, how the body processes elritercept, and the effects of elritercept on anemia when taken with or without ruxolitinib The study will also check on how safe elritercept is and how well it is tolerated.

DETAILED DESCRIPTION:
Elritercept is an investigational therapeutic protein designed to increase red blood cell and platelet production by inhibiting the signaling of a subset of the transforming growth factor beta (TGF-ß) family of proteins to promote hematopoiesis. It is being developed for the treatment of low blood cell counts, or cytopenias including anemia and thrombocytopenia in participants with Myelodysplastic Syndrome (MDS) and Myelofibrosis (MF).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national and local study participant privacy regulations.
2. In the opinion of the Investigator, the participant is able and willing to comply with the requirements of the protocol (e.g., all study procedures, return for follow-up visits).
3. Male or female greater than equal to (≥)18 years of age, at the time of signing informed consent.
4. Eastern Cooperative Oncology Group (ECOG) performance score lesser than equal to (≤)2.
5. Life expectancy ≥12 months per Investigator assessment.
6. Confirmed diagnosis of primary myelofibrosis (PMF) (prefibrotic or overtly fibrotic) according to the 2016 World Health Organization (WHO) criteria, post-polycythemia vera myelofibrosis (PV MF), or post-essential thrombocythemia myelofibrosis (ET MF) according to the 2008 International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) criteria.
7. Anemia, defined as:

   1. Having received ≥6 units of RBC transfusion for Hgb ≤8.5 g/dL in the 12 weeks prior to the planned C1D1, including ≥1 unit of RBC transfusion in the 28 days prior to C1D1; or
   2. Having ≥3 evaluable Hgb measurements at less than (<)10.0 g/dL including ≥1 evaluable Hgb measurement assessed 8 to 13 weeks prior to C1D1. Participants receiving RBC transfusions but not meeting criterion "a." may enroll under criterion "b." following the below parameters:

      * All pre-transfusion Hgb values (defined as a Hgb assessed within the 3 days prior to a transfusion) should be recorded, and ≥1 pre-transfusion Hgb value is required.
      * Hgb values collected within the 28 days following a transfusion will not be considered evaluable unless qualifying as a pre-transfusion Hgb; in cases where multiple transfusions are given in succession due to poor Hgb response, only the first pre-transfusion Hgb will be considered evaluable.
8. Arm-specific criteria:

   Arms 1A and 2A:
   1. Previously treated with JAK inhibitor(s) and, per the Investigator, discontinued due to one of the following reasons:

      * Relapsed disease following treatment with JAK inhibitor(s)
      * Refractory to treatment with JAK inhibitor(s)
      * Intolerance to treatment with JAK inhibitor(s)
      * Participant no longer met risk/benefit ratio to continue JAK inhibitor(s) OR
      * Participant with prognostic score of intermediate-1 or higher per Dynamic International Prognostic Scoring System (DIPSS) and is ineligible for JAK inhibitor(s) in the opinion of the Investigator
   2. Participants previously treated with JAK inhibitor(s) must have discontinued JAK inhibitor therapy ≥8 weeks before C1D1

   Arms 1B and 2B:
   1. Has been receiving ruxolitinib prescribed for a diagnosis of PMF (prefibrotic or overtly fibrotic), post-PV MF, or post-ET MF for ≥8 weeks prior to C1D1 and on a stable dose for ≥4 weeks prior to C1D1. In Arm 2B only, at least 10 participants should have been on ruxolitinib for <6 months prior to C1D1.
   2. Meets ≥1 of the following criteria in the opinion of the Investigator:

      * Current ruxolitinib treatment is considered to be providing insufficient control of the disease
      * The participant's cytopenias are limiting the participant's ruxolitinib dose intensity
      * The participant's disease is symptomatic and warrants additional therapy

   Arm 2C (Brazil only):
   1. No prior treatment with JAK inhibitor(s) and no access to JAK inhibitor therapy as determined by the Investigator
   2. Spleen volume ≥ 450 cubic centimeter (cm^3) as assessed by CT or MRI collected during the pretreatment period and/or
   3. Myelofibrosis Symptom Assessment Form Total Symptom Score (MF-SAF-TSS) meeting at least one of the following criteria during the pretreatment period:

      * 2 symptoms with average score ≥ 3
      * Average total symptom score ≥ 10
9. Females of childbearing potential and sexually active males must agree to use highly effective methods of contraception as described in the protocol.

Exclusion Criteria:

Medical History:

1. Active infection requiring parenteral antibiotic therapy within 28 days prior to C1D1 or oral antibiotics within 14 days of C1D1. Prophylactic antibiotics and/or antifungals for neutropenia are allowed.
2. Presence of the following cardiac conditions:

   1. New York Heart Association Class 3 or 4 heart failure
   2. QTcF (QT interval corrected by Fridericia's formula) >500 milliseconds (msec) on the screening or C1D1 electrocardiogram (ECG; mean of 3 measurements)
   3. Uncontrolled clinically significant arrhythmia (participants with rate-controlled atrial fibrillation are not excluded)
   4. Acute myocardial infarction or unstable angina pectoris ≤6 months prior to C1D1
3. Body mass index (BMI) ≥40 kilograms per meter square (kg/m^2).
4. Presence of uncontrolled hypertension, defined as systolic blood pressure ≥160 millimeters of mercury (mmHg) or diastolic blood pressure ≥100 mmHg despite adequate treatment.
5. History of drug or alcohol abuse (as defined by the Investigator) within the past 2 years.
6. History of stroke, deep venous thrombosis, or arterial embolism within 6 months prior to C1D1.
7. Major surgery within 28 days prior to C1D1. Participants must have completely recovered from any previous surgery prior to C1D1 in the opinion of the Investigator.
8. Known positive for human immunodeficiency virus (HIV), active infectious hepatitis B with positive viral load (hepatitis B virus [HBV] deoxyribonucleic acid [DNA]), or active infectious hepatitis C with positive viral load (hepatitis C virus [HCV] ribonucleic acid [RNA]). Participants without a known positive history of HIV, HBV, and/or HCV do not require further testing, unless testing is mandated per local guidelines.
9. Any malignancy other than PMF, post-ET MF, or post-PV MF that has not been in remission and/or has required systemic therapy including radiation, chemotherapy, hormonal therapy, or biologic therapy, within 1 year prior to C1D1. In situ cancers, squamous cell and basal cell carcinomas, and monoclonal gammopathy of unclear significance are allowed at the discretion of the Investigator.
10. History of solid organ or hematological transplantation.
11. History of severe allergic or anaphylactic reaction(s) or hypersensitivity to recombinant proteins or excipients in the investigational drug, or ruxolitinib for participants enrolling in Arm 1B or 2B.
12. Diagnosis of hemolytic anemia, active bleeding, hemoglobinopathies, or congenital disorders as a cause of the participant's anemia.
13. History of intracranial hemorrhage (any grade).
14. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 bleeding events within the 3 months prior to C1D1.
15. Receipt of an RBC or platelet transfusion for any reason(s) or combination of reasons other than underlying MF within the 12 weeks prior to C1D1. If a participant requires a transfusion for an unanticipated reason during the Pretreatment Period, a prolonged screening period may be considered after discussion with the Medical Monitor.

    Treatment History:
16. Prior treatment with luspatercept, sotatercept, or other commercially available or investigational transforming growth factor-beta (TGF-β) inhibitors (all arms).
17. Treatment within 28 days prior to C1D1 with:

    1. Erythropoiesis-stimulating agent (ESA)
    2. Granulocyte colony-stimulating factor (G-CSF)
    3. Granulocyte-macrophage colony-stimulating factor (GM-CSF)
    4. Thrombopoietin (TPO) agonists
    5. Immunomodulator imide drugs (IMiDs) (e.g., thalidomide, pomalidomide, lenalidomide)
    6. Interferon
    7. Hydroxyurea
    8. Steroids at doses exceeding corticosteroid equivalent of 10 mg/day prednisone
18. Newly initiated iron chelation therapy within the 8 weeks prior to C1D1. Stable doses of iron chelators are allowed if prescribed per label.
19. Vitamin B12 and/or folate therapy initiated within 4 weeks before randomization. Participants on stable replacement doses for ≥4 weeks and without concurrent vitamin B12 or folate deficiency are allowed.
20. Treatment with another investigational drug or device or approved therapy for the treatment of MF or anemia in MF ≤28 days prior to C1D1, or, if the half-life of the previous product is known, within 5 times the half-life prior to C1D1, whichever is longer.
21. For Arms 1B and 2B (participants receiving ruxolitinib), initiation of treatment with strong cytochrome P450 (CYP)3A4 inhibitors within 2 weeks prior to C1D1. Participants receiving CYP3A4 inhibitors/inducers as concomitant therapy with ruxolitinib in accordance with ruxolitinib local prescribing information may continue to receive such therapies in this study.

    Laboratory Exclusions (during screening):
22. Bone marrow aspirate blast percentage >5 percent (%)

    a. In the event of a non-evaluable pretreatment bone marrow aspirate expected to be due to marrow fibrosis, participants may be enrolled without bone marrow aspirate blast percentage data if all other eligibility criteria are met. Historical bone marrow data may be requested to support confirmation of diagnosis.
23. Peripheral blood blast percentage ≥10%
24. Platelet count <25 × 10^9 per liter (10^9/)L or >450 × 10^9/L
25. Persistent Hgb <7 g/dL despite RBC transfusions
26. Transferrin saturation <15%
27. Ferritin <50 nanograms per mililiters (ng/mL)
28. Folate <4.5 nanomoles per liter (nmol/L) (<2.0 picograms per liter (pg/L))
29. Vitamin B12 <148 picomoles per liter (pmol/L) (<200 picograms per milliliter (pg/mL))
30. Estimated glomerular filtration rate <30 milliliters per minute per 1.73 square meter (mL/min/1.73 m^2) (as determined by the Chronic Kidney Disease Epidemiology Collaboration equation)
31. Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >3 × upper limit of normal (ULN)
32. Total bilirubin >2 × ULN
33. International normalized ratio (INR) >1.2 × ULN, unless participant is receiving anticoagulation, in which instance the INR must fall within the participant's designated therapeutic range.

    Miscellaneous:
34. Pregnant or lactating females.
35. Any other condition not specifically noted above that, in the opinion of the Investigator or Sponsor, would preclude the participant from participating in the study.
36. Participants who are investigational site staff members directly involved in the conduct of the study and their immediate family members, site staff members otherwise supervised by the Investigator, or participants who are Keros or contract research organization (CRO) employees directly involved in the conduct of the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Adverse Events (AEs), Dose Limiting Toxicities (DLTs), Severe Adverse Events (AEs) and Serious Adverse Events (SAEs) | From signing of the informed consent form (ICF) through 30 days after the last dose of study drug (approximately 8 years)
  AE:any untoward medical occurrence (MO) in clinical study participant administered medicinal product not necessarily having causal relationship with treatment.Severe AE medically significant AE but not immediately life-threatening;may result in hospitalization/ prolonged hospital stay;disability.SAE:any untoward MO that,at any dose results in death,is life-threatening,requires in-patient hospitalization/ prolongation of existing hospitalization,results in persistent or significant disability/incapacity,is congenital anomaly/birth defect,is medically important event.DLT: any following safety events-death,Grade 4 neutropenia/ thrombocytopenia >7 days,Grade 3 thrombocytopenia with bleeding,Neutropenic fever,assessments meeting Hy's law,Grade ≥3 nonhematologic treatment-emergent adverse events(TEAEs),elevated hemoglobin(Hgb)/ platelet count requiring dose modification, other safety event considered by Safety Review Committee(SRC) to be significant to warrant categorization as DLT.
Part 2 and Long-Term Extension: Number of Participants with Adverse Events (AEs), Severe AEs and SAEs | From signing of the ICF through 30 days after the last dose of study drug, (approximately 8 years)
  An AE is defined as any untoward medical occurrence in a clinical study participant administered a medicinal product that does not necessarily have a causal relationship with this treatment. Severe AE is defined as an AE which is medically significant but not immediately life-threatening; may result in hospitalization or prolonged hospital stay; disabling. An SAE is any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event.

SECONDARY OUTCOMES:
Percentage of Participants with Progression to Acute Myeloid Leukemia (AML) | From signing of the ICF through 30 days after the last dose of study drug, (approximately 8 years)
Percentage of Participants with Progression to Accelerated MF | From signing of the ICF through 30 days after the last dose of study drug, (approximately 8 years)
Percentage of Participants with Red Blood Cell (RBC) Transfusion Independence Over a Period of ≥12 Consecutive Weeks | Up to Week 24
  Participants with anemia requiring RBC transfusions will be assessed for this outcome measure.
Percentage of Participants with RBC Transfusions From Baseline Over a Period of ≥12 Consecutive Weeks | Up to Week 24
  Participants with anemia requiring RBC transfusions will be assessed for this outcome measure and percentage of participants with ≥50% decrease in number of RBC transfusions will be represented.
Percentage of Participants with Mean Haemoglobin (Hgb) Increase From Baseline Over a Period of ≥12 Consecutive Weeks | Up to Week 24
  Participants with transfusion-independence will be assessed for this outcome measure for mean Hgb ≥1.5 grams per deciliter (g/dL) and ≥2.0 g/dL.
Percentage of Participants with Improvement in the Myelofibrosis Symptom Assessment Form Version 4.0 Total Symptom Score (MF-SAF(v4.0)-TSS) From Baseline at Week 24 | Week 24
  Percentage of participants with MF-SAF(v4.0)-TSS of ≥50% will be presented for this assessment. MF-SAF v4.0 captures participant self-report of 7 core MF symptoms (this includes fatigue, night sweats, itching, abdominal discomfort, pain under ribs on left side, early satiety, and bone pain) over the past 7 days. Response options range from 0 (absent) to 10 (worst imaginable). The TSS is computed by averaging the individual item responses and multiplying by 7 for a weekly total score ranging from 0 to 70. Higher scores represent higher symptom burden.
Percentage of Participants with Decrease in Spleen Volume From Baseline as Measured by Computed Tomography/Magnetic Resonance Imaging (CT/MRI) at Week 24 | Week 24
  Percentage of participants with decrease in spleen volume of ≥35% will be presented for this outcome measure.
Plasma Concentrations of Elritercept | Within 2 hours before administration of elritercept at multiple timepoints up to 8 weeks after the end of treatment
Maximum Observed Serum Concentration (Cmax) of Elritercept | Within 2 hours before administration of elritercept at multiple timepoints up to 8 weeks after the end of treatment
Time to Maximum Observed Concentration (Tmax) of Elritercept | Within 2 hours before administration of elritercept at multiple timepoints up to 8 weeks after the end of treatment
Area Under the Concentration-time Curve From Time 0 to the Time of Last Quantifiable Concentration (AUC0-last) of Elritercept | Through Cycle 1 (each cycle=28 days)
Minimum Observed Serum Concentration (Cmin) of Elritercept | Within 2 hours before administration of elritercept at multiple timepoints up to 8 weeks after the end of treatment
Accumulation Rate (Rac) of Elritercept | Within 2 hours before administration of elritercept at multiple timepoints up to 8 weeks after the end of treatment
Change From Baseline in Red Cell Parameters | At multiple timepoints from pre-treatment period up to 8 weeks after end of treatment
  The red cell parameters including reticulocyte count, Hgb, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), and reticulocyte cell Hgb will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (46):
- Australia (6):
  - Concord Hospital, Concord, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Flinders Medical Centre, Woodville South, South Australia
  - St. Vincents Hospital Melbourne, Fitzroy, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Ballarat Oncology & Haematology Service, Wendouree, Victoria
- Brazil (6):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - IMV-Pesquisa Cardiologica Sociedade Simples, Porto Alegre
  - Albert Einstein Sociedade Beneficente Israelita Brasiliera, São Paulo
  - Hospital Beneficencia Portuguesa de Sao Paulo, São Paulo
  - Hospital Das Clinicas Da Faculdade de Medicina Da U S P, São Paulo
  - Instituto de Ensino e Pesquisas Sao Lucas, São Paulo
- France (6):
  - CHU Amiens - Hopital Sud, Amiens
  - Hopital Morvan, Brest
  - Hopital Prive Sevigne, Cesson-Sévigné
  - Centre Hospitalier Lyon Sud, Lyon
  - Institut de Cancerologie du Gard, Nîmes
  - Hopital de la Source - CHR Orleans, Orléans
- Italy (12):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino, Genova
  - ASST Grande Ospedale Metropolitano Niguarda, Niguarda Cancer Center, Milan
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Milan
  - Arcispedale S. Maria Nuova Azienda Ospedaliera di Reggio Emilia, Reggio Emilia
  - Azienda Ospedaliera Universitaria Policlinico Umberto I, Roma
  - Azienda Socio Sanitaria Territoriale Sette Laghi, Varese
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- South Korea (4):
  - Gachon University Gil Medical Center, Incheon
  - Samsung Medical Center, Seoul
  - Seoul St. Marys Hospital, The Catholic University of Korea, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
- Spain (7):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital QuironSalud de Zaragoza, Zaragoza
- United Kingdom (5):
  - United Lincolnshire Hospitals NHS Trust - Pilgrim Hospital, Boston
  - St James Hospital,Leeds, Leeds
  - Guys Hospital, London
  - Hammersmith Hospital, London
  - University College London, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.